CLINICAL TRIAL: NCT05169177
Title: Radio-opaque Contrast Agents for Liver Cancer Targeting With KIM During Radiation Therapy
Acronym: ROCK-RT
Status: Recruiting | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: Calvary Mater Newcastle, Australia (Other); Western Sydney Local Health District (Other); Austin Health (Other Government); Peter MacCallum Cancer Centre, Australia (Other); Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: IX-2020-DS-ROCKRT
Record Dates: First submitted 2021-12-08; First posted 2021-12-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Liver Neoplasm
Keywords: Radiation Therapy; Stereotactic Ablative Body Radiation Therapy; SABR; Kilovoltage intrafraction monitoring; Radio opaque contrast
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study will investigate the properties of image files standardly collected during radiation therapy treatment in a cross-section of liver cancer patients who received stereotactic ablative body radiation therapy (SABR) after trans-catheter arterial chemo emobilisation (TACE). Specifically, it will determine whether the radio-opaque contrast agents in the image files can be detected by tumour-tracking software (KIM).

DETAILED DESCRIPTION:
* Sites will collect image files from the Cancer Radiation Therapy Systems and the medical records of eligible participants. For patient who do not have implanted markers, research personnel (a radiation oncologist, medical physicist or radiation therapist) will manually outline the visible contrast mass. This outline is considered the 'ground truth' of the location of the contrast mass. To ensure its accuracy, the ground truth contrast mass location will be checked by research personnel from another study site.
* Image and ground truth data collected from 80% of participants will be used by University of Sydney researchers to develop the KIM algorithm to detect and track the radio-opaque contrast agents with sufficient robustness to provide justification for the prospective use of KIM as a real-time image guided radiation therapy tool for liver cancer patients.
* The developed KIM software will be applied by site Medical Physicist(s) to the treatment imaging data from the remaining 20% of participants the images. Tumour positions produced by KIM will be compared with a 'ground truth' manual delineation.

ELIGIBILITY:
Inclusion Criteria:

* Received or will receive stereotactic ablative body radiotherapy (SABR) treatment for liver cancer at a participating site.
* Received a radio-opaque contrast agent (e.g. Lipiodol™ or DC Bead LUMI™) that is visible on the radiation treatment planning CT scan
* The radio-opaque contrast agent mass is or will be within the x-ray imaging field of view during the CBCT scan and any planned intra-fraction imaging. Note that there is no requirement of the distance between the contrast agent mass and the treated tumour as the goal of the study is the contrast agent mass tracking.
* Provides written informed consent (prospectively recruited) or meets criteria for waiving of the requirement for consent (retrospectively recruited)

Exclusion Criteria:

* Less than 18 years of age
* Minimum image dataset is not available
* Image dataset is not in a compatible format

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had or will have SABR for liver cancer following TACE chemotherapy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of images that have contrast mass detection by software | 2 weeks
  Proportion of images in which kilovoltage intrafraction monitoring software detects contrast agent mass on CBCT and intra-treatment images
Average difference between software and ground truth measure | 2 weeks
  Average difference (mm) of location of contrast mass detection on CBCT and treatment images by KIM software compared to the ground truth in each of the horizontal and vertical directions.
Standard deviation of difference between software and ground truth measure | 2 weeks
  Standard deviation difference (mm) of location of contrast mass detection on CBCT and treatment images by KIM software compared to the ground truth in each of the horizontal and vertical directions.

SECONDARY OUTCOMES:
Modelling of patient or treatment features that contributed to the success or failure of the KIM method | 2 weeks
  Using the KIM success rate (primary hypothesis) and patient CT imaging features (contrast agent density, size, shape and location, patient size etc) a generalised linear model, or appropriate alternative, will be used to identity univariate and multivariate patient or treatment features that contributed to the success or failure of the KIM method. Selected features will be identified and developed into a model. If the model predicts the likelihood of KIM success in at least 85% of the patients then the study will be deemed to have achieved the hypothesis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, PhD, Study Chair — University of Sydney
Locations (5):
- Australia (5):
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Austin Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
After study completion, de-identified (non-coded, non-re-identifiable) data may be shared with researchers for further scientific research. Information about data sharing will be provided to study participants in the Patient Information Sheet.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study analyses and publications are complete.
Access Criteria: Data stored at the university: In order to download / decompress the stored, de-identified data, participating researchers will agree to the terms of use for the data, including: (i) that the data are not to be published or otherwise redistributed without the express consent of the original investigator(s) and (ii) that the data are forbidden to be used for any commercial purpose.
  Data stored at an external repository: de-identified study data may be provided to an eternal research data repository, archive or register so that it may be made publicly available for other scientific research. Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board, under a Materials Transfer Agreement with the university.

REFERENCES:
- [Derived] Plant N, Mylonas A, Sengupta C, Nguyen DT, Silvester S, Pryor D, Greer P, Lee YYD, Ramachandran P, Seshadri V, Trada Y, Khor R, Wang T, Hardcastle N, Keall P. Radio-opaque contrast agents for liver cancer targeting with KIM during radiation therapy (ROCK-RT): an observational feasibility study. Radiat Oncol. 2024 Oct 8;19(1):139. doi: 10.1186/s13014-024-02524-4. PMID 39380004